CLINICAL TRIAL: NCT01320722
Title: Modifiable Effectors of Renin System Activation: Treatment Evaluation (MODERATE)
Brief Title: Study of Vitamin D and Uric Acid Lowering on Kidney and Blood Vessel Function
Acronym: MODERATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, John P. Forman, INSTRUCTOR IN MEDICINE, BRIGHAM AND WOMEN'S HOSPITAL, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-P-002049; 1R01HL105440 (NIH)
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Renal Function; Endothelial Function; Blood Pressure; Overweight; Obesity
Keywords: renin angiotensin system; vitamin D; uric acid; allopurinol; probenecid; endothelial function
MeSH Terms: conditions — Overweight; Obesity | interventions — Ergocalciferols; Vitamin D; Probenecid; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Vitamin D (Experimental): Vitamin D ergocalciferol 50,000 unit soft gel capsule once per week for 8 weeks.
  Interventions: Drug: Vitamin D ergocalciferol
- Probenecid (Experimental): Probenecid 500 mg tablet once per day for 4 weeks, then either 500 mg tablet once per day for 4 weeks or 1000 mg once per day for 4 weeks (8 weeks total).
  Interventions: Drug: Probenecid
- Allopurinol (Experimental): Allopurinol 300 mg tablet once per day for 4 weeks then either 300 mg once per day or 600 mg once per day for 4 weeks (8 weeks total).
  Interventions: Drug: Allopurinol
- Placebo- Vitamin D (Placebo Comparator): Placebo soft gel once per week for 8 weeks.
  Interventions: Drug: Placebo
- Placebo- Uric Acid (Placebo Comparator): Placebo tablet once per day for 4 weeks then twice per day for 4 weeks (eight weeks total).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D ergocalciferol — 50,000 unit soft gel capsule once per week for 8 weeks
  Other Names: Vitamin D
  Arms: Vitamin D
Drug: Probenecid — 500 mg tablet once per day for 4 weeks, then either 500 mg tablet once per day for 4 weeks or 1000 mg once per day for 4 weeks (8 weeks total)
  Arms: Probenecid
Drug: Allopurinol — 300 mg tablet once per day for 4 weeks then either 300 mg once per day or 600 mg once per day for 4 weeks (8 weeks total)
  Arms: Allopurinol
Drug: Placebo — Placebo soft gel once per week for 8 weeks
  Arms: Placebo- Vitamin D
Drug: Placebo — Placebo tablet once per day for 4 weeks then twice per day for 4 weeks (eight weeks total)
  Arms: Placebo- Uric Acid

SUMMARY:
The investigators hypothesize that, among non-hypertensive overweight and obese individuals, treatment of vitamin D deficiency and lowering uric acid concentrations (by either xanthine oxidase inhibition or increased renal excretion) will attenuate renin angiotensin system (RAS) activation, improve endothelial function, and lower blood pressure.

DETAILED DESCRIPTION:
We have demonstrated that lower levels of 25-hydroxyvitamin D (25[OH]D) and higher concentrations of uric acid are both potentially modifiable factors that are independently associated with an increased risk of developing hypertension (high blood pressure) in humans. Other investigators have shown that vitamin D supplementation, or lowering uric acid with allopurinol, may reduce blood pressure. Animal experiments suggest that activation of both the systemic and local kidney-specific renin angiotensin systems (RAS) may be the principal mechanism linking 25(OH)D and uric acid with hypertension. In human parallels to these animal studies, we have shown in cross-sectional analyses that non-hypertensive individuals with lower 25(OH)D and higher uric acid levels have increased activation of their systemic and kidney-specific RAS, independent of other factors. However, whether vitamin D supplementation or uric acid lowering attenuates RAS activation has never been demonstrated in humans. Both lower 25(OH)D and higher uric acid concentrations are also associated with endothelial dysfunction in humans, and endothelial function may modulate the RAS and provide an alternate mechanism for the development of hypertension. It remains unclear, however, whether an intervention to increase 25(OH)D or decrease uric acid levels among non-hypertensive adults improves endothelial function; furthermore, it is unknown whether treatment of these individuals would lower blood pressure. Determining whether treatment of 25(OH)D and uric acid concentrations, per se, can attenuate RAS activation, improve endothelial function, and lower blood pressure among nonhypertensive individuals is critically important, with implications stretching beyond hypertension prevention, since RAS activation, endothelial dysfunction, and blood pressure are also implicated in the pathology of cardiovascular and chronic kidney disease. Individuals who are overweight and obese (two-thirds of US adults) represent an important population who are known to have lower 25(OH)D levels, higher uric acid concentrations, activation of the RAS, endothelial dysfunction, and an increased risk of hypertension, cardiovascular disease, and chronic kidney disease. Interestingly, our preliminary data demonstrate that among overweight and obese individuals with normal 25(OH)D or low uric acid levels, adiposity is no longer associated with activation of the RAS, suggesting that low 25(OH)D and high uric acid concentrations might be mediators of the adverse consequences of overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* 25(OH)D < 20 ng/mL OR Uric acid ≥ 5 mg/dL
* Age ≥ 18, ≤ 75 years
* Body Mass Index (BMI) ≥ 25 kg/m^2

Exclusion Criteria:

* Hypertension, or on BP-lowering medicine
* Diabetes
* Coronary Heart Disease
* estimated glomerular filtration rate (EGFR) <60 mL/min
* Kidney stones
* Active cancer (except non-melanoma skin cancer)
* Pregnant
* Taking vitamin D supplements and unwilling to stop
* Osteoporosis
* Hypo- or hypercalcemia
* Hypo- or hyperphosphatemia
* Known allergy to angiotensin-converting enzyme (ACE)-inhibitors
* Taking medication for hyperuricemia
* Gout, anemia, cirrhosis, active/chronic hepatitis, abnormal aspartate aminotransferase (AST), alanine aminotransferase (ALT) or total bilirubin levels, or anemia
* Known allergy to either allopurinol or probenecid
* Current use of didanosine, azothioprine, methotrexate, ketoprofen, ketorolac, mycophenolate, or ACE-inhibitors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2011-03; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Forman, MD, MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D | Placebo- Vitamin D | Probenecid | Allopurinol | Placebo- Uric Acid
Started | 46 | 47 | 47 | 49 | 53
Received Intervention | 43 | 45 | 46 | 48 | 51
Completed | 43 | 41 | 40 | 35 | 45
Not Completed | 3 | 6 | 7 | 14 | 8
Not completed — Did not Receive Intervention | 3 | 2 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 3
Not completed — Not Available for the 8 Week Visit | 0 | 3 | 0 | 0 | 0
Not completed — Participant Developed a Rash | 0 | 0 | 2 | 1 | 1
Not completed — Non-compliant with Medication | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 6 | 0
Not completed — Not Compliant with Study Procedures | 0 | 0 | 0 | 4 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0
Not completed — Started an Exclusionary Medication | 0 | 0 | 0 | 0 | 1
Not completed — Withdrew due to Health Condition | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo- Vitamin D | Probenecid | Allopurinol | Placebo- Uric Acid | Total
Number analyzed (Participants) | 46 | 47 | 47 | 49 | 53 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All randomized participants in the Vitamin D arms.
  years
    number analyzed (Participants) | 46 | 47 | 0 | 0 | 0 | 93
    (all) | 39 (13) | 35 (11) |  |  |  | 37 (12.3)
Age, Continuous [Mean (Standard Deviation); unit: years] — All randomized participants. Population: All randomized participants in the Uric Acid arms.
  years
    number analyzed (Participants) | 0 | 0 | 47 | 49 | 53 | 149
    (all) |  |  | 37 (14) | 43 (12.5) | 41 (14) | 41 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 23 | 24 | 28 | 137
  Male | 15 | 16 | 24 | 25 | 25 | 105
Change in Renal Plasma Flow (RPF) in Response to Captopril [Vitamin D] [Mean (Standard Deviation); unit: milliliters(mL)/minute(min) per 1.73 m^2] — An 8 milligrams (mg)/kilogram(kg) loading dose of para-aminohippuric acid (PAH) was given, immediately followed by a continuous PAH infusion at 12 mg/minute. After 60 minutes a single dose of 25 mg of captopril was administered. Three pre-captopril measurements and three post-captopril measurements of RPF were made. RPF was normalized to body surface area of 1.73 meters squared (m^2). The change in RPF was calculated as post-captopril RPF- pre-captopril RPF. Population: All randomized participants in the Vitamin D arms with data available for RPF.
  milliliters(mL)/minute(min) per 1.73 m^2
    number analyzed (Participants) | 43 | 41 | 0 | 0 | 0 | 84
    (all) | 33.9 (56.1) | 37.3 (46.9) |  |  |  | 35.6 (50.0)
Change in RPF in Response to Captopril [Uric Acid] [Mean (Standard Deviation); unit: mL/min per 1.73 m^2] — An 8 milligrams (mg)/kilogram(kg) loading dose of para-aminohippuric acid (PAH) was given, immediately followed by a continuous PAH infusion at 12 mg/minute. After 60 minutes a single dose of 25 mg of captopril was administered. Three pre-captopril measurements and three post-captopril measurements of RPF were made. RPF was normalized to body surface area of 1.73 meters squared (m^2). The change in RPF was calculated as post-captopril RPF- pre-captopril RPF. Population: All randomized participants in the Uric Acid arms with data available for RPF.
  mL/min per 1.73 m^2
    number analyzed (Participants) | 0 | 0 | 40 | 45 | 53 | 138
    (all) |  |  | 38 (46.0) | 41 (32.2) | 30 (35.5) | 36.3 (38.7)
Plasma Renin Activity (PRA) [Vitamin D] [Mean (Standard Deviation); unit: nanograms (ng)/mL per hour] — Population: All randomized participants in the Vitamin D arms with data available for PRA.
  nanograms (ng)/mL per hour
    number analyzed (Participants) | 43 | 41 | 0 | 0 | 0 | 84
    (all) | 0.34 (0.37) | 0.42 (0.44) |  |  |  | 0.38 (0.40)
Plasma Renin Activity (PRA) [Uric Acid] [Mean (Standard Deviation); unit: ng/mL] — Population: All randomized participants in the Uric Acid arms with data available for PRA.
  ng/mL
    number analyzed (Participants) | 0 | 0 | 39 | 35 | 43 | 117
    (all) |  |  | 0.3 (0.52) | 0.3 (0.33) | 0.2 (0.33) | 0.27 (0.40)
Angiotensin II Concentration (ATII) [Vitamin D] [Mean (Standard Deviation); unit: picogram(pg)/mL] — Population: All randomized participants in the Vitamin D arms with data available for ATII.
  picogram(pg)/mL
    number analyzed (Participants) | 43 | 41 | 0 | 0 | 0 | 84
    (all) | 19.9 (5.9) | 19.9 (4.5) |  |  |  | 19.9 (5.0)
Angiotensin II Concentration (ATII) [Uric Acid] [Mean (Standard Deviation); unit: pg/mL] — Population: All randomized participants in the Uric Acid arms with data available for ATII.
  pg/mL
    number analyzed (Participants) | 0 | 0 | 40 | 34 | 45 | 119
    (all) |  |  | 19.6 (5.0) | 18.9 (4.0) | 18.8 (4.8) | 19.1 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Renal Plasma Flow (RPF) in Response to Captopril in High Sodium Balance [Vitamin D]
Description: Change in RPF in response to captopril is a measure of the vasodilator effect from inhibiting angiotensin II (AngII)- mediated vascular tone and therefore the degree of kidney specific Renin Angiotensin System (RAS) activity. Participants consumed a high sodium diet 3 days prior to the test. Following an 8 hour fast, participants remained in a supine (lying down) position and had an intravenous (IV) catheter inserted in each arm, one for infusion and one for blood collection. An 8 milligrams (mg)/kilogram(kg) loading dose of para-aminohippuric acid (PAH) was given, immediately followed by a continuous PAH infusion at 12 mg/minute. After 60 minutes a single dose of 25 mg of captopril was administered. Three pre-captopril measurements and three post-captopril measurements of RPF were made. RPF was normalized to body surface area of 1.73 meters squared (m^2). The change in RPF was calculated as post-captopril RPF- pre-captopril RPF.
Time Frame: Week 8 (pre and post captopril)
Population: All randomized enrolled participants included in the analysis.
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Vitamin D | Placebo- Vitamin D
Number analyzed (Participants) | 43 | 41
mL/min per 1.73 m^2 | 35.7 (47.7) | 35.9 (26.2)
Statistical Analysis 1: Comparison: Vitamin D vs Placebo- Vitamin D; Week 8; Test type: Superiority; p = 0.72, Repeated Measures Analysis

2. Primary Outcome: Plasma Renin Activity (PRA) [Vitamin D]
Description: PRA is a measure of systemic renin angiotensin system (RAS) activation. Blood was collected and plasma PRA was analyzed using a competitive binding radioimmunoassay (RIA) laboratory test.
Time Frame: Week 8
Population: All randomized enrolled participants included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL per hour
Arm/Group | Vitamin D | Placebo- Vitamin D
Number analyzed (Participants) | 43 | 41
ng/mL per hour | 0.36 (0.44) | 0.44 (0.8)
Statistical Analysis 1: Comparison: Vitamin D vs Placebo- Vitamin D; Week 8; Test type: Superiority; p = 0.77, t-test, 2 sided — Statistical significance was set for P>0.05

3. Primary Outcome: Angiotensin II (ATII) Concentration [Vitamin D]
Description: ATII concentration is a measure of systemic renin angiotensin system (RAS) activation. Blood was collected and plasma ATII was analyzed using a double-antibody radioimmunoassay (RIA) laboratory test.
Time Frame: Week 8
Population: All randomized enrolled participants included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vitamin D | Placebo- Vitamin D
Number analyzed (Participants) | 43 | 41
pg/mL | 19.5 (4.4) | 19.7 (7.1)
Statistical Analysis 1: Comparison: Vitamin D vs Placebo- Vitamin D; Week 8; Test type: Superiority; p = 0.57, t-test, 2 sided — Statistical significance was set for P>0.05

4. Primary Outcome: Change in Renal Plasma Flow (RPF) Response to Captopril in High Sodium Balance [Uric Acid]
Description: RPF in response to captopril iis a measure of the vasodilator effect from inhibiting angiotensin II (AngII)- mediated vascular tone and therefore the degree of kidney specific Renin Angiotensin System (RAS) activity. Participants consumed a high sodium diet 3 days prior to the test. Following an 8 hour fast, participants remained in a supine (lying down) position and had an intravenous (IV) catheter inserted in each arm, one for infusion and one for blood collection. An 8 milligrams (mg)/kilogram(kg) loading dose of para-aminohippuric acid (PAH) was given, immediately followed by a continuous PAH infusion at 12 mg/minute. After 60 minutes a single dose of 25 mg of captopril was administered. Three pre-captopril measurements and three post-captopril measurements of RPF were made. RPF was normalized to body surface area of 1.73 meters squared (m^2). The change in RPF was calculated as post-captopril RPF- pre-captopril RPF.
Time Frame: Week 8 (pre and post captopril)
Population: All randomized enrolled participants with data available for analysis.
Measure: Median (Inter-Quartile Range); unit: mL/min per 1.73 m^2
Arm/Group | Probenecid | Allopurinol | Placebo- Uric Acid
Number analyzed (Participants) | 40 | 34 | 45
mL/min per 1.73 m^2 | 33 [12 to 72] | 36 [17 to 55] | 30 [-1 to 48]
Statistical Analysis 1: Comparison: Probenecid vs Placebo- Uric Acid; Test type: Superiority; p = 0.8, Repeated Measures Analysis
Statistical Analysis 2: Comparison: Allopurinol vs Placebo- Uric Acid; Test type: Superiority; p = 0.6, Repeated Measures Analysis

5. Primary Outcome: Plasma Renin Activity (PRA) [Uric Acid]
Description: as for outcome 2
Time Frame: Week 8
Population: All randomized enrolled participants with data available for analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mL per hour
Arm/Group | Probenecid | Allopurinol | Placebo- Uric Acid
Number analyzed (Participants) | 40 | 33 | 44
ng/mL per hour | 0.4 [0.2 to 0.7] | 0.3 [0.2 to 0.5] | 0.2 [0.1 to 0.6]
Statistical Analysis 1: Comparison: Probenecid vs Placebo- Uric Acid; Test type: Superiority; p = 0.6, Repeated Measures Analysis
Statistical Analysis 2: Comparison: Allopurinol vs Placebo- Uric Acid; Test type: Superiority; p = 0.7, Repeated Measures Analysis

6. Primary Outcome: Angiotensin II (ATII) Concentration [Uric Acid]
Description: as for outcome 3
Time Frame: Week 8
Population: All randomized enrolled participants with data available for analysis.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Probenecid | Allopurinol | Placebo- Uric Acid
Number analyzed (Participants) | 39 | 34 | 45
pg/mL | 20.3 [18.5 to 22.7] | 21.4 [18.2 to 24.4] | 19.1 [17.0 to 21.5]
Statistical Analysis 1: Comparison: Probenecid vs Placebo- Uric Acid; Test type: Superiority; p = 0.3, Repeated Measures Analysis
Statistical Analysis 2: Comparison: Allopurinol vs Placebo- Uric Acid; Test type: Superiority; p = 0.1, Repeated Measures Analysis

7. Secondary Outcome: Change in Endothelium-Dependent Vasodilation (EDV)
Description: Endothelial function was assessed by EDV using brachial artery ultrasonography. Measurements of brachial artery diameter were made under basal conditions and reactive hyperemia following ischaemic stimulus. A blood pressure cuff on the forearm was pumped up for 5 minutes then released. Images were taken at baseline and after reactive hyperemia (increased blood flow). The maximum diameter was determined by the investigator. Change in EDV was expressed as a percent of brachial luminal diameter calculated as post-ischaemic brachial artery diameter - pre-ischaemic brachial artery diameter/pre-ischaemic brachial artery diameter * 100.
Time Frame: Baseline and Week 8 (pre and post ischaemic stimulus)
Population: All randomized enrolled participants.
Measure: Mean (Standard Deviation); unit: percent of brachial luminal diameter
Arm/Group | Vitamin D | Placebo- Vitamin D | Probenecid | Allopurinol | Placebo- Uric Acid
Number analyzed (Participants) | 46 | 47 | 47 | 49 | 53
percent of brachial luminal diameter
  Baseline | 6.3 (3.6) | 7.9 (4.7) | 7.4 (5.1) | 7.6 (6.0) | 6.5 (3.8)
  Week 8 | 6.1 (4.6) | 6.8 (4.7) | 8.3 (5.1) | 6.2 (4.8) | 7.1 (4.9)
Statistical Analysis 1: Comparison: Vitamin D vs Placebo- Vitamin D; Week 8; Test type: Superiority or Other; p = 0.35, t-test, 2 sided; Statistical significance was set for a 2-tailed P <0.05
Statistical Analysis 2: Comparison: Probenecid vs Placebo- Uric Acid; Week 8; Test type: Superiority; p = 0.7, t-test, 2 sided — Statistical significance was set for a 2-tailed P <0.05
Statistical Analysis 3: Comparison: Allopurinol vs Placebo- Uric Acid; Week 8; Test type: Superiority; p = 0.06, t-test, 2 sided — Statistical significance was set for a 2-tailed P <0.05

8. Secondary Outcome: Mean 24-Hour Ambulatory Blood Pressure (ABP)
Description: A 24-hour mean ambulatory blood pressure was monitored using a 24 hour ABP device. The ABP device is a small box that is worn on the belt or pant/skirt line with a line that connect under the clothing to the cuff on the upper arm. Blood Pressure was recorded every 30 minutes during the day and every 60 minutes during the night for 24 hours.
Time Frame: Baseline and Week 8
Population: All randomized enrolled participants with complete 24-hour ABP data available for analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vitamin D | Placebo- Vitamin D | Probenecid | Allopurinol | Placebo- Uric Acid
Number analyzed (Participants) | 29 | 27 | 25 | 27 | 30
mmHg
  Overall Systolic Blood Pressure (SBP), Baseline | 120.4 (10.2) | 123.7 (7.6) | 126.9 (10.2) | 124.1 (8.8) | 122.4 (9.7)
  Overall Diastolic Blood Pressure (DBP), Baseline | 71.6 (6.4) | 73.7 (5.8) | 73.3 (7.8) | 72.1 (7.1) | 71.9 (7.4)
  Awake SBP, Baseline | 122.4 (10.9) | 126.4 (7.4) | 130.0 (9.2) | 126.7 (8.4) | 125.5 (9.0)
  Asleep SBP, Baseline | 113.9 (11.0) | 116.5 (8.7) | 119.2 (12.4) | 117.1 (10.0) | 113.9 (12.2)
  Overall SBP, Week 8 | 121.6 (8.3) | 124.7 (9.6) | 125.2 (9.1) | 123.7 (9.4) | 122.9 (9.5)
  Overall DBP, Week 8 | 72.0 (5.6) | 74.7 (7.2) | 73.8 (6.9) | 72.0 (6.5) | 72.6 (6.2)
  Awake SBP, Week 8 | 124.2 (9.1) | 127.6 (9.2) | 128.1 (9.3) | 125.1 (9.6) | 124.9 (10.1)
  Asleep SBP, Week 8 | 114.7 (8.1) | 117.4 (11.4) | 116.2 (9.6) | 118.6 (11.7) | 116.2 (10.5)
Statistical Analysis 1: Comparison: Vitamin D vs Placebo- Vitamin D; Overall SBP; Test type: Superiority; p = 0.92, Repeated Measures Analysis — Statistical significance was set for P>0.05
Statistical Analysis 2: Comparison: Vitamin D vs Placebo- Vitamin D; Overall DBP; Test type: Superiority; p = 0.64, Repeated Measures Analysis — Statistical significance was set for P>0.05
Statistical Analysis 3: Comparison: Vitamin D vs Placebo- Vitamin D; Awake SBP; Test type: Superiority; p = 0.80, Repeated Measures Analysis — Statistical significance was set for P>0.05
Statistical Analysis 4: Comparison: Vitamin D vs Placebo- Vitamin D; Asleep SBP at Week 8; Test type: Superiority; p = 0.97, Repeated Measures Analysis — Statistical significance was set for P>0.05
Statistical Analysis 5: Comparison: Probenecid vs Placebo- Uric Acid; Overall SBP; Test type: Superiority; p = 0.34, Repeated Measures Analysis
Statistical Analysis 6: Comparison: Probenecid vs Placebo- Uric Acid; Overall DBP; Test type: Superiority; p = 0.59, Repeated Measures Analysi
Statistical Analysis 7: Comparison: Probenecid vs Placebo- Uric Acid; Awake SBF; Test type: Superiority; p = 0.57, Repeated Measures Analysis
Statistical Analysis 8: Comparison: Probenecid vs Placebo- Uric Acid; Asleep SBP; Test type: Superiority; p = 0.08, Repeated Measures Analysis
Statistical Analysis 9: Comparison: Allopurinol vs Placebo- Uric Acid; Overall SBP; Test type: Superiority; p = 0.59, Repeated Measures Analysis
Statistical Analysis 10: Comparison: Allopurinol; Test type: Superiority; p = 0.53, Repeated Measures Analysis
Statistical Analysis 11: Comparison: Allopurinol vs Placebo- Uric Acid; Awake SBP; Test type: Superiority; p = 0.55, Repeated Measures Analysis
Statistical Analysis 12: Comparison: Allopurinol vs Placebo- Uric Acid; Asleep SBP; Test type: Superiority; p = 0.80, Repeated Measures Analysis

9. Secondary Outcome: Mean 24-Hour Ambulatory Blood Pressure (ABP) Nocturnal Dipping
Description: A 24-hour mean ambulatory blood pressure was monitored using a 24 hour ABP device. The ABP device is a small box that is worn on the belt or pant/skirt line with a line that connect under the clothing to the cuff on the upper arm. Blood Pressure was recorded every 30 minutes during the day and every 60 minutes during the night for 24 hours. Nocturnal dipping is the percent change lower between the daytime and nighttime values.
Time Frame: Baseline and Week 8
Population: All randomized enrolled participants with complete 24-hour ABP data available for analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vitamin D | Placebo- Vitamin D | Probenecid | Allopurinol | Placebo- Uric Acid
Number analyzed (Participants) | 29 | 27 | 25 | 27 | 30
percent change
  Baseline | 7.3 (6.3) | 7.8 (5.1) | 8.4 (6.8) | 7.5 (5.3) | 9.4 (6.2)
  Week 8 | 7.5 (5.7) | 8.1 (6.0) | 9.2 (6.1) | 5.2 (7.1) | 6.9 (6.2)
Statistical Analysis 1: Comparison: Vitamin D vs Placebo- Vitamin D; Test type: Superiority; p = 0.98, Repeated Measures Analysis
Statistical Analysis 2: Comparison: Probenecid vs Placebo- Uric Acid; Test type: Superiority; p = 0.07, Repeated Measures Analysis
Statistical Analysis 3: Comparison: Allopurinol vs Placebo- Uric Acid; Test type: Superiority; p = 0.97, Repeated Measures Analysis

ADVERSE EVENTS:
Description: All randomized participants who received study intervention.
Arm/Group | Vitamin D | Placebo- Vitamin D | Probenecid | Allopurinol | Placebo- Uric Acid
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/45 | 4/46 | 6/48 | 2/51
Other Adverse Events (participants affected / at risk) | 5/43 | 6/45 | 16/46 | 36/48 | 25/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D (N=43) | Placebo- Vitamin D (N=45) | Probenecid (N=46) | Allopurinol (N=48) | Placebo- Uric Acid (N=51)
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 1
Elevated creatinine (Investigations) | 0 | 0 | 1 | 3 | 0
Elevated liver enzymes (Investigations) | 0 | 0 | 0 | 3 | 1
Decreased hematocrit (Investigations) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin D (N=43) | Placebo- Vitamin D (N=45) | Probenecid (N=46) | Allopurinol (N=48) | Placebo- Uric Acid (N=51)
Abdominal discomfort (Gastrointestinal disorders) | 4 | 4 | 1 | 6 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Elevated phosphorus (Investigations) | 0 | 1 | 0 | 0 | 0
Elevated potassium (Investigations) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 3 | 2 | 2
Fatigue (General disorders) | 0 | 0 | 4 | 4 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 3
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Tingling in extremities (General disorders) | 0 | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 4
Altered taste (General disorders) | 0 | 0 | 0 | 3 | 2
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Heartburn (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Transient shortness of breath (General disorders) | 0 | 0 | 0 | 2 | 0
Transient nose bleed (General disorders) | 0 | 0 | 0 | 1 | 0
Transient facial swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Unusual reaction to bee sting (General disorders) | 0 | 0 | 0 | 0 | 1
Sleepiness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Difficulty sleeping (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sensitivity to touch (Nervous system disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes